CLINICAL TRIAL: NCT06480006
Title: Evaluation of the Validity and Reliability of the BETY-Biopsychosocial Questionnaire in Individuals With Coronary Artery Disease
Brief Title: Validity and Reliability of the BETY-Biopsychosocial Questionnaire in Individuals With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Professor, Hacettepe University
Other Study IDs: SBA 24/353
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Validity; Reliability
Keywords: BETY- Biopsychosocial Questionnaire (BETY-BQ); Validity; Reliability; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scales for biopsychosocial assessment of coronary artery disease patients are limited. The aim of this study was to evaluate the validity and reliability of the Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire (BETY-BQ) in patients with CAD.

DETAILED DESCRIPTION:
Ischaemic heart disease, also called coronary heart disease (CHD), is associated with obstruction of epicardial coronary arteries and inadequate blood supply to the myocardium, usually caused by atherosclerosis, which may result in the development of obstructive plaque called atheroma. Imbalance in lipid accumulation and chronic inflammation of the vessel wall are considered to be the main causes of atherosclerosis. Multiple pathophysiological mechanisms can cause CAD. The most common atherosclerotic epicardial coronary artery occlusion is the most common. However, one third of patients may not have significant epicardial disease and often have microvascular disease as the underlying pathophysiology. The Cognitive Exercise Therapy Approach (BETY) is an exercise-based biopsychosocial approach that has been ongoing for 14 years, in which individuals of all ages with various rheumatic diseases participate in group exercises three days a week. A biopsychosocial scale called BETY-Biopsychosocial Questionnaire (BETY-BQ) was created in line with the feedback received from patients who participated in this group for many years and the changes that occurred in them. The patients mentioned that the existing scales did not measure the changes that occurred in them as a result of their participation in the BETY group for many years. As a result, the answers given by the patients to the question "So what changes have you experienced?" were collected. Reverse expressions of these sentences were created and the scale item pool was formed by determining the complaints when they did not receive treatment, expert opinions were taken and the validity of the scale was finalised with rheumatic patients. BETY-BQ includes items that provide information about pain, sociability, mood, sexuality, functionality and sleep quality.

Demographic characteristics and clinical information were recorded: Participants' age, diagnosis, gender, education level, occupation, marital status, body weight, height, body mass index, background, family history, monthly income level, lifestyle characteristics (smoking, exercise habits) will be recorded. In addition, clinical history of CAD, number of daily medications and drug groups, and additional chronic diseases will be questioned.

Cardiovascular Disease Risk Scoring: SCORE2. The SCORE risk scoring was developed by analysing data from studies in 12 European countries, with more than 200,000 participants, approximately 3 million annual follow-ups and more than 7,000 cardiovascular deaths. In the SCORE table, which has a high applicability in primary care, 10-year CVD event risk is determined by using age, gender, total cholesterol, smoking status and blood pressure values. All atherosclerotic deaths (not only deaths due to CAD) are taken into account in the risk calculation and stroke-related deaths can be separated from CAD-related deaths when desired. Studies in the SCORE database have shown that HDL-cholesterol may have a significant effect on risk calculation. When HDL-cholesterol values are included in the SCORE tables, it is seen that the risk changes at all risk levels, at all ages and genders. The updated SCORE algorithm, SCORE2, incorporates the effect of the non-HDL-cholesterol value and estimates an individual's 10-year risk of fatal and non-fatal CVD events (myocardial infarction, stroke) in apparently healthy people aged 40-69 years with risk factors. SCORE2 and SCORE2-OP are calibrated according to four country clusters (low, intermediate, high and very high CVD risk) grouped according to national CVD mortality rates published by WHO. Turkey is in the group of high-risk countries. The risk calculated according to the SCORE system is considered low risk if <1%, medium risk if 1-4%, high risk if 5-9%, and very high risk if 10% and above. According to the SCORE2 system, those under the age of 50 are considered to be at low-moderate risk if <2.5%, high risk if 2.5%-7.5%, and very high risk if 7.5% and above. In those over 50 years of age, <5% is considered low-moderate risk, 5-10% is considered high risk, and 10% and above is considered very high risk.

Quality of life assessment: Short Form-36 (Short Form-36, SF-36) will be used. The scale consists of 36 items, which are grouped into 8 subscales: physical function (10 items), role limitations related to physical function (4 items), role limitations related to emotional problems (3 items), energy/vitality (4 items), mental health (5 items), social function (2 items), pain (2 items) and general health perception (5 items). The assessment covers the last 4 weeks. Each subgroup is scored within itself. Scoring is in the range of 0-100 and the higher the score, the better the quality of life. In addition, 2 summary scales, physical component scale (PCS) and mental component scale (MCS), can be made. The physical component scale consists of physical function, role limitations related to physical functions, pain and general health perception subgroups, while the mental component scale consists of role limitations related to emotional problems, energy/vitality, mental health and social function subgroups.

Assessment of anxiety and depression: The Hospital Anxiety and Depression Scale (HADS) was developed by Zigmond and Snaith (1983). The scale consists of 14 items. Seven of these items measure anxiety and the other seven items measure depression symptoms. The items in the scale are evaluated with a 4-point Likert scale and are based on a scoring system between 0-3. According to the scoring, 0-1 is considered as not ill, 2 as borderline ill, and 2-3 as severely ill. It is also observed that the scores obtained from the scale are not affected by physical diseases. The aim of the scale is not to make a diagnosis, but to measure the psychological state of the patients and to take necessary precautions.

Assessment of Biopsychosocial Characteristics: Cognitive Exercise Therapy Approach- Biopsychosocial Scale (BETY-BQ) will be used to evaluate individuals in terms of biopsychosocial aspects. The scale has sub-dimensions that determine the biopsychosocial characteristics of individuals. It includes pain, functionality, mood, sociability, sexuality and sleep parameters. BETY-BQ is a 5-point Likert-type scale consisting of 30 items in total. When the items of the scale are examined in detail, items 1,2,3,4,5 define the Pain sub-dimension, items 6,7,8,9,10,11,12,26,28 define the Functionality sub-dimension, items 13,14,15,16,16,17,18,18,19,20,21,22 define the Emotional State sub-dimension, items 23,24,25 define the Sociability sub-dimension, items 27,29 define the Sexuality sub-dimension and item 30 defines the Sleep sub-dimension. It offers a measurement between 0-120 values as scoring. The sub-dimensions score range is Pain 0-20, Functionality 0-36, Emotional State 0-40, Sociability 0-12, Sexuality 0-8, Sleep 0-4. It gives the opportunity to evaluate individuals with both sub-dimensions and total score. High scores indicate low quality of life and poor biopsychosocial status.

Kinesiophobia Assessment: Patients' kinesiophobia will be assessed with the Turkish version of the Tampa Kinesiophobia Rating for the Heart (KTKD), a valid and reliable scale developed for cardiac diseases. The KTKD assesses the subjective evaluation of kinesiophobia in relation to cardiac conditions. These statements are made on a four-point Likert scale ranging from "strongly disagree" (score 1) to "strongly agree" (score 4). The scale consists of four subgroups including exercise avoidance, fear of injury, perceived danger of cardiac problems and dysfunction. The 11-question Turkish version of the scale has been shown to be valid and reliable in patients with heart failure and PH, and written permission was obtained for its use in this study.

Assessment of Disease Specific Quality of Life: It will be evaluated with the Seattle Angina Questionnaire (SAQ). SAQ is a disease-specific scale developed to evaluate functional capacity in patients with angina. SAQ has five subscales (physical function, angina stability, angina frequency, treatment satisfaction and perception of quality of life). It consists of 19 items. Each item is answered using a 5 or 6-point Likert scale. Each subscale is scored from 0 (worst health status) to 100 (best health status).

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-80
* Volunteering to participate in the research
* Having coronary artery disease (CAD)
* Having no problem in reading and/or understanding the scales and being able to cooperate with the tests.

Exclusion Criteria:

* Active infection,
* No history of myocardial infarction, angina pectoris, percutaneous transluminal coronary angioplasty or bypass surgery in file records and medical history,
* Having a neurological disease or other clinical diagnosis that may affect cognitive status.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 years who were diagnosed with coronary artery disease (CAD) in the Department of Internal Medicine, Division of General Internal Medicine, Hacettepe University Hospital and who volunteered to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Biopsychosocial Characteristics | One Year
  Assessment of Biopsychosocial Characteristics: BETY-Biopsychosocial Questionnaire:It offers a measurement between 0-120 values as scoring. The sub-dimensions score range is Pain 0-20, Functionality 0-36, Emotional State 0-40, Sociability 0-12, Sexuality 0-8, Sleep 0-4. It gives the opportunity to evaluate individuals with both sub-dimensions and total score. A high score indicates low quality of life and poor biopsychosocial status.

SECONDARY OUTCOMES:
Quality of life | One Year
  Short Form-36 questionnaire: The scale consists of 36 items, which are grouped into 8 subscales: physical functioning (10 items), role limitations related to physical functioning (4 items), role limitations related to emotional problems (3 items), energy/vitality (4 items), mental health (5 items), social functioning (2 items), pain (2 items) and general health perception (5 items). The assessment covers the last 4 weeks. Each subgroup is scored on its own. Scoring is in the range of 0-100 and the higher the score, the better the quality of life.
Kinesiophobia | One Year
  Turkish version of the Tampa Kinesiophobia Rating for the Heart (KTKD): The scale uses a 4-point Likert scale (1= Strongly disagree, 4= Strongly agree). After reversing items 4, 8, 12 and 16, a total score is calculated. The person receives a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Anxiety and Depression | One Year
  The Hospital Anxiety and Depression Scale (HADS):The scale consists of 14 items. Seven of these items measure anxiety symptoms and the other seven items measure depression symptoms. The items in the scale are evaluated on a 4-point Likert scale and are based on a scoring system between 0-3. According to the scoring, 0-1 is considered as not ill, 2 as borderline ill, and 2-3 as severely ill.
Cardiovascular Disease Risk Scoring | One Year
  SCORE2: According to the SCORE2 system, those under 50 years of age are considered low-moderate risk if <2.5%, high risk if 2.5%-7.5%, and very high risk if 7.5% and above. In those over 50 years of age, <5% is considered low-moderate risk, 5-10% is considered high risk, and 10% and above is considered very high risk.
Functional Status | One Year
  Seattle Angina Questionnaire (SAQ): SAQ with its five subscales (physical function, angina stability, angina frequency, treatment satisfaction and perception of quality of life) It consists of 19 items. Each item is answered using a 5 or 6-point Likert scale. Each subscale is scored from 0 (worst health) to 100 (best health).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided